CLINICAL TRIAL: NCT00470977
Title: Treatment of Exudative and Vasogenic Chorioretinal Diseases Including Variants of AMD and Other CNV Related Maculopathy With Intravitreal Injection of Lucentis (Ranibizumab Injection)
Brief Title: Treatment of Exudative and Vasogenic Chorioretinal Diseases Including Variants of AMD and Other CNV Related Maculopathy
Acronym: FVF4140S
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Joan, Lawrence A. Yannuzzi, M.D., Manhattan Eye, Ear & Throat Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol: FVF4140S
Record Dates: First submitted 2007-05-04; First posted 2007-05-08 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Coats' Disease; Idiopathic Retinal Telangiectasia; Retinal Angiomatous Proliferation; Polypoidal Choroidal Vasculopathy; Pseudoxanthoma Elasticum; Pathological Myopia; Multi-focal Choroiditis; Rubeosis Iridis; Von Hippel Lindau Disease; BEST VITELLIFORM MACULAR DYSTROPHY, MULTIFOCAL (Disorder)
MeSH Terms: conditions — Retinal Telangiectasis; Polypoidal Choroidal Vasculopathy; Pseudoxanthoma Elasticum; Myopia, Degenerative; von Hippel-Lindau Disease; Vitelliform Macular Dystrophy | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- (Ranibizumab) Lucentis (Experimental): (Ranibizumab)Lucentis 0.5%
  Interventions: Drug: ranibizumab injection (0.5 mg)

INTERVENTIONS:
Drug: ranibizumab injection (0.5 mg) — ranibizumab 10mg mg/ml. , 0.3ml/vial, 0.05 ml./injection intravitreally for 3months then prn for the next 21 months.
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of intravitreal injections of ranibizumab in the treatment of AMD variants and other choroidal neovascularization (CNV) related conditions (Coats' disease, idiopathic perifoveal telangiectasia, retinal angiomatous proliferation, polypoidal vasculopathy, pseudoxanthoma elasticum, pathological myopia, multi-focal choroiditis, rubeosis iridis) using the incidence and severity of adverse events.

Limited forms of treatment are available that limit the loss of visual acuity. However, the patients may not have any substantial improvement in acuity or function. Therefore there remains a significant unmet need for therapeutic options managing the neovascularization and its consequences.

Lucentis (ranibizumab) injection will be considered as an attempt to control the growth of the abnormal vessels because of evidence suggesting that angiogenic factors, such as vascular endothelial growth factor (VEGF), play a role in the pathogenesis of neovascular non-AMD conditions.

The rationale for the study design is as follows:

A 0.5 mg dose of Lucentis (ranibizumab), a commercially available preparation that is Food and Drug Administration (FDA) approved and labeled for intravitreal injection use for neovascular (wet) age-related macular degeneration will be used.

In AMD variants and other CNV related conditions, vascular endothelial growth factor (VEGF) plays a role in the pathogenesis as in neovascular AMD.

Intravitreal injection of ranibizumab delivers maximal concentration of the antibody fragment to the vitreous cavity with minimal systemic exposure. The dosing schedule, based on considerations of the half-life and the clinical response in patients with neovascularization suggests that a 1-month interval is optimal.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

1. Ability to provide written informed consent and comply with study assessments for the full duration of the study
2. Age > 18 years
3. Clinical diagnosis of the following conditions: Coats' disease, idiopathic perifoveal telangiectasia, retinal angiomatous proliferation, polypoidal vasculopathy, pseudoxanthoma elasticum, pathological myopia, multi-focal choroiditis, rubeosis iridis.
4. Visual acuity of 20/40 to 20/320 in the study eye on the ETDRS visual acuity chart.
5. Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

1. Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy is initiated
2. Participation in another simultaneous medical investigation or trial
3. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
4. Patients who have undergone intraocular surgery within the last 2 months.
5. Patient participating in any other investigational drug study.
6. Use of an investigational drug or treatment related or unrelated to the patient's condition within 30 days prior to receipt of study medication (verteporfin, pegaptanib, or other AMD therapy in the study eye)
7. Patient treated with systemic anti-VEGF or pro-VEGF agents within 3 months before enrollment.
8. Previous treatment (in either eye) with intravitreal or intravenously administered Avastin (bevacizumab).
9. Inability to obtain photographs to document CNV (including difficulty with venous access).
10. Patient with a known adverse reaction to fluorescein dye.
11. Patient has a history of any medical condition which would preclude scheduled visits or completion of the study.
12. Patient has had insertion of scleral buckle in the study eye
13. Patient has received radiation treatment.
14. Aphakia or absence of the posterior capsule in the study eye. Previous violation of the posterior capsule in the study eye is also excluded unless as a result of yttrium aluminum garnet (YAG) posterior capsulotomy in association with posterior chamber lens implantation.
15. Pregnancy (positive pregnancy test) or lactation.
16. Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an intrauterine device (IUD), or contraceptive hormone implant or patch.
17. History of glaucoma filtering surgery in the study eye.
18. Concurrent use of more than two therapies for glaucoma.
19. Uncontrolled glaucoma in the study eye (defined as intraocular pressure > 30 mm Hg despite treatment with anti-glaucoma medication)
20. Inability to comply with study or follow-up procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of intravitreal injections of ranibizumab in the treatment of non-AMD variants and other CNV related conditions | 24 months

SECONDARY OUTCOMES:
Mean change in central retinal thickness as measured by OCT at month 12 compared to baseline | 24 months
Change in leakage area seen during fluorescein angiography at month 12 as compared with baseline | 24 months
Number of additional injections required following the initial 3 injections | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Yannuzzi, MD, Principal Investigator — LuEsther T. Mertz Retinal Research Center
Locations (2):
- United States (2):
  - Lenox Hill Hospital/Manhattan Eye Ear and Throat Institute, New York, New York
  - Lenox Hill Hospital/Manhattan Eye, Ear & Throat Institute, New York, New York